CLINICAL TRIAL: NCT01945944
Title: Nebulized Hypertonic Saline for Mechanically Ventilated Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Steven Shein, Attending Physician, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-13-11
Record Dates: First submitted 2013-09-12; First posted 2013-09-19 (Estimated); Results first posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-05

CONDITIONS: Respiratory Failure
Keywords: pediatric; mucolytic; respiratory failure; atelectasis; hypertonic saline
MeSH Terms: conditions — Respiratory Insufficiency; Pulmonary Atelectasis | interventions — Saline Solution, Hypertonic; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo (0.9% saline), 3mL every 6 hrs for up to 7 days
  Interventions: Drug: Placebo (0.9% saline)
- Hypertonic Saline (Experimental): Hypertonic saline (3%), 3mL every 6hrs for up to 7 days
  Interventions: Drug: Hypertonic saline (3%)

INTERVENTIONS:
Drug: Hypertonic saline (3%) — 3mL of HTS given via nebulizer every 6hrs
  Other Names: 3% saline
  Arms: Hypertonic Saline
Drug: Placebo (0.9% saline) — 3mL of normal saline given via nebulizer every 6hrs
  Other Names: normal saline
  Arms: Placebo

SUMMARY:
Children who need to be on a ventilator often have thick secretions/mucus in their lungs. These secretions can obstruct the breathing tube and their windpipe, which can worsen lung function and prolong the need for the ventilator. Hypertonic saline is a medicine that is used to thin out secretions in patients with cystic fibrosis (and other conditions). We hypothesize that having children on a ventilator inhale this medication will shorten the amount of time that they need to be on the ventilator.

DETAILED DESCRIPTION:
Recent pediatric data shows that less than 80% of children mechanically ventilated for ≥ 96 hours survived to PICU discharge, while 100% of children mechanically ventilated for < 96 hours survived to PICU discharge. Interventions that decrease duration of mechanical ventilation may improve outcome by limiting ventilator-induced lung injury, sedative medication usage and ventilator-associated pneumonia. Obstructive airway secretions may prolong mechanical ventilation by causing atelectasis and endotracheal tube obstruction, with resultant cardio-respiratory instability. Nebulized hypertonic saline (HTS) is used to decrease mucus viscosity and increase mucociliary clearance in patients with diseases such as cystic fibrosis and bronchiolitis, and has been used to enhance airway clearance in mechanically ventilated children. Administering nebulized HTS to mechanically ventilated children may facilitate airway clearance and shorten mechanical ventilation.

In a randomized study of children < 2 years old following cardiac surgery, patients given dornase, another mucolytic agent, had a significantly decreased duration of mechanical ventilation versus those given saline placebo (52 hrs vs. 82 hrs). HTS may be even more effective, as mechanically ventilated newborns with persistent atelectasis had more improvement in radiographic findings and oxygen saturation when randomized to receive hypertonic saline compared to those randomized to receive dornase. This may be because dornase may only be effective in patients with leukocytes or bacterial present in tracheal aspirates, while HTS may be effective in all ventilated patients. Further study of the impact of prophylactic mucolytic therapy on the duration of mechanical ventilation in children is warranted.

ELIGIBILITY:
Inclusion Criteria:

* invasive mechanical ventilation of < 12 hrs duration prior to enrollment
* expected duration of mechanical ventilation of > 48hrs from enrollment
* age < 18yo

Exclusion Criteria:

* inclusion in another clinical study
* cystic fibrosis
* status asthmaticus
* pulmonary hemorrhage/contusion
* home O2 use
* home non-invasive positive pressure (CPAP/BiPAP) ventilation use
* pre-existing tracheostomy
* prescription of mucolytic medication by primary clinical team
* allergy to inhaled saline/hypertonic saline or albuterol

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Shein, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- Rainbow Babies and Children's Hospital (of Univ. Hospitals Case Med. Center), Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Payen V, Jouvet P, Lacroix J, Ducruet T, Gauvin F. Risk factors associated with increased length of mechanical ventilation in children. Pediatr Crit Care Med. 2012 Mar;13(2):152-7. doi: 10.1097/PCC.0b013e3182257a24. PMID 21760567
- [Background] Riethmueller J, Borth-Bruhns T, Kumpf M, Vonthein R, Wiskirchen J, Stern M, Hofbeck M, Baden W. Recombinant human deoxyribonuclease shortens ventilation time in young, mechanically ventilated children. Pediatr Pulmonol. 2006 Jan;41(1):61-6. doi: 10.1002/ppul.20298. PMID 16265663
- [Background] Dilmen U, Karagol BS, Oguz SS. Nebulized hypertonic saline and recombinant human DNase in the treatment of pulmonary atelectasis in newborns. Pediatr Int. 2011 Jun;53(3):328-31. doi: 10.1111/j.1442-200X.2010.03245.x. PMID 20831650
- [Background] Prodhan P, Greenberg B, Bhutta AT, Hyde C, Vankatesan A, Imamura M, Jaquiss RD, Dyamenahalli U. Recombinant human deoxyribonuclease improves atelectasis in mechanically ventilated children with cardiac disease. Congenit Heart Dis. 2009 May-Jun;4(3):166-73. doi: 10.1111/j.1747-0803.2009.00289.x. PMID 19489944
- [Background] Zhang L, Mendoza-Sassi RA, Wainwright C, Klassen TP. Nebulized hypertonic saline solution for acute bronchiolitis in infants. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD006458. doi: 10.1002/14651858.CD006458.pub2. PMID 18843717
- [Background] Rosenfeld M, Ratjen F, Brumback L, Daniel S, Rowbotham R, McNamara S, Johnson R, Kronmal R, Davis SD; ISIS Study Group. Inhaled hypertonic saline in infants and children younger than 6 years with cystic fibrosis: the ISIS randomized controlled trial. JAMA. 2012 Jun 6;307(21):2269-77. doi: 10.1001/jama.2012.5214. PMID 22610452
- [Background] Elkins MR, Robinson M, Rose BR, Harbour C, Moriarty CP, Marks GB, Belousova EG, Xuan W, Bye PT; National Hypertonic Saline in Cystic Fibrosis (NHSCF) Study Group. A controlled trial of long-term inhaled hypertonic saline in patients with cystic fibrosis. N Engl J Med. 2006 Jan 19;354(3):229-40. doi: 10.1056/NEJMoa043900. PMID 16421364
- [Background] Altunhan H, Annagur A, Pekcan S, Ors R, Koc H. Comparing the efficacy of nebulizer recombinant human DNase and hypertonic saline as monotherapy and combined treatment in the treatment of persistent atelectasis in mechanically ventilated newborns. Pediatr Int. 2012 Feb;54(1):131-6. doi: 10.1111/j.1442-200X.2011.03519.x. PMID 22114907
- [Background] Youness HA, Mathews K, Elya MK, Kinasewitz GT, Keddissi JI. Dornase alpha compared to hypertonic saline for lung atelectasis in critically ill patients. J Aerosol Med Pulm Drug Deliv. 2012 Dec;25(6):342-8. doi: 10.1089/jamp.2011.0954. Epub 2012 Mar 13. PMID 22413805

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo (0.9% saline), 3mL every 6 hrs for up to 7 days
  Placebo (0.9% saline)
- Hypertonic Saline: Hypertonic saline (3%), 3mL every 6hrs for up to 7 days
  Hypertonic saline (3%)
Period: Overall Study
Arm/Group | Placebo | Hypertonic Saline
Started | 9 | 9
Completed | 8 | 6
Not Completed | 1 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Hypertonic Saline | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Median (Inter-Quartile Range); unit: weeks] | 26 [3.1 to 174.2] | 12.7 [5.6 to 32.6] | 17.9 [5.1 to 44.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 6 | 7 | 13
Race/Ethnicity, Customized [Number; unit: participants]
  African-American | 4 | 5 | 9
  Caucasian | 5 | 3 | 8
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18
PEEP (positive end-expiratory pressure) [Median (Inter-Quartile Range); unit: cm-H20] | 5 [5 to 6] | 7 [6.5 to 8] | 6 [5 to 7]

OUTCOME MEASURES:

1. Primary Outcome: Duration of Mechanical Ventilation
Time Frame: typically 4 days - 2 weeks
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Placebo | Hypertonic Saline
Number analyzed (Participants) | 9 | 9
hours | 129.5 [74.4 to 146.1] | 208.1 [136.3 to 319.8]

2. Secondary Outcome: Atelectasis
Description: using chest x ray score. The score measures the amount of lung collapse ("atelectasis") observed on a chest x-ray. For each of the 5 lung lobes, 1 point is given for linear atelectasis, 2 points for sub-segmental atelectasis and 3 points for lobar atelectasis. The range is 0-15 points, with higher scores reflecting more severe lung collapse.
Time Frame: during mechanical ventilation (typically 4 days - 2 weeks)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Hypertonic Saline
Number analyzed (Participants) | 9 | 9
units on a scale | 4.67 [3.92 to 6] | 4 [2.33 to 5.83]

3. Secondary Outcome: Wheezing
Description: as dichotomous outcome (yes/no) following drug administration
Time Frame: during mechanical ventilation (typically 4 days - 2 weeks)
Measure: Number; unit: percentage of drug doses w/ wheezing
Arm/Group | Placebo | Hypertonic Saline
Number analyzed (Participants) | 9 | 9
percentage of drug doses w/ wheezing | 3 | 1

4. Secondary Outcome: ICU Length of Stay
Time Frame: during hospitalization (typically 4 days - 2 weeks)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Hypertonic Saline
Number analyzed (Participants) | 9 | 9
days | 8 [6 to 12.5] | 12 [9 to 17]

5. Secondary Outcome: Hospital Length of Stay
Time Frame: during hospitalization (typically 4 days - 2 weeks)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Hypertonic Saline
Number analyzed (Participants) | 9 | 9
days | 15 [9 to 22.5] | 17 [16 to 22.5]

6. Secondary Outcome: Change in Serum Sodium From Baseline
Description: The baseline sodium was the last level measured prior to study initiation, typically within 24hrs of study initiation. The change in blood sodium level was calculated as the difference between the mean post-enrollment sodium level during ICU care and the sodium level at enrollment.
Time Frame: during hospitalization (typically 4 days - 2 weeks)
Measure: Median (Inter-Quartile Range); unit: mEq/L
Arm/Group | Placebo | Hypertonic Saline
Number analyzed (Participants) | 9 | 9
mEq/L | 1 [-0.9 to 6.7] | -1.5 [-4.1 to 7.1]

7. Secondary Outcome: Dynamic Compliance
Description: measured in ml/cm H20/kg using parameters on mechanical ventilator
Time Frame: during mechanical ventilation (typically 4 days - 2 weeks)
Measure: Median (Inter-Quartile Range); unit: mL/kg/cm-H20
Arm/Group | Placebo | Hypertonic Saline
Number analyzed (Participants) | 9 | 9
mL/kg/cm-H20 | 6.52 [4.21 to 8.14] | 4.47 [2.94 to 7]

8. Secondary Outcome: Oxygenation
Description: SaO2/FiO2. This is a measure of how will the lungs are providing oxygen to the body. Higher ratios reflect better lung function.
Time Frame: during mechanical ventilation (typically 4 days - 2 weeks)
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Placebo | Hypertonic Saline
Number analyzed (Participants) | 9 | 9
ratio | 239 [196 to 280] | 188 [162 to 239]

9. Secondary Outcome: Dead Space
Description: in % of tidal volume, using parameters on mechanical ventilator. Dead space is a measure of how much of the lung is not able to move air into and out of the body. Higher levels of dead space reflect higher levels of lung dysfunction.
Time Frame: during mechanical ventilation (typically 4 days - 2 weeks)
Measure: Median (Inter-Quartile Range); unit: percentage of lung volume
Arm/Group | Placebo | Hypertonic Saline
Number analyzed (Participants) | 9 | 9
percentage of lung volume | 29 [20 to 37] | 37 [26 to 45]

ADVERSE EVENTS:
Arm/Group | Placebo | Hypertonic Saline
Serious Adverse Events (participants affected / at risk) | 0/9 | 2/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | Hypertonic Saline (N=9)
Desaturation (oxygen) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
As shown above, baseline lung function (as measured by PEEP) was worse in the treatment (HTS) group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No